CLINICAL TRIAL: NCT06301360
Title: How Much Does the Therapist Matter in Internet Based Emotional Awareness and Expression Therapy (I-EAET) for Functional Somatic Disorder? A Randomised Controlled Trial of I-EAET With and Without Therapist Support
Brief Title: Internet Based Emotional Awareness and Expression Therapy for Functional Somatic Disorder With and Without Therapist Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Maroti (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor-Investigator, Daniel Maroti, PhD, principal investigator, Stockholm University
Organization: Stockholm University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOSMOS2 2023-04956-01
Record Dates: First submitted 2024-02-27; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Functional Somatic Disorder; Somatic Symptom Disorder; Functional Somatic Syndromes
Keywords: Internet based interventions; EAET; Psychodynamic therapy

STUDY DESIGN:
Intervention Model Description: RCT with two treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-EAET with therapist support (Experimental): I-EAET is a 10 week treatment intervention combining principles from emotion focused therapies and neuroscience. Main components include psychoeducation on the body-mind connection, anxiety regulation with self-compassion exercises and different techniques for emotional exposure and processing. Participants have help from a therapist giving feedback.
  Interventions: Behavioral: Internet based Emotional Awareness and Expression Therapy (I-EAET)
- I-EAET without therapist support (Active Comparator): I-EAET is a 10 week treatment intervention combining principles from emotion focused therapies and neuroscience. Main components include psychoeducation on the body-mind connection, anxiety regulation with self-compassion exercises and different techniques for emotional exposure and processing. Participants works on their own and have only technical support.
  Interventions: Behavioral: Internet based Emotional Awareness and Expression Therapy (I-EAET)

INTERVENTIONS:
Behavioral: Internet based Emotional Awareness and Expression Therapy (I-EAET) — In I-EAET with therapist support, the therapist and participants communicate asynchronous using written messages. The therapist gives feedback each week on home-work assignments and is available on demand for support.
  In I-EAET without therapist support, the participants works with home-work assignments on their own and only have technical support.

SUMMARY:
Functional somatic syndromes (e.g. irritable bowel syndrome, fibromyalgia) and medically unexplained symptoms (e.g. chronic primary pain) are very common in primary care. These patients make 14 times more doctor visits than the general population, but describe themselves as less satisfied with the care they receive. Although Region Stockholm in Sweden recently developed care flows based on 'step up' care for the most common patient groups in primary care, patients with functional or medically unexplained symptoms are not mentioned.

Short-term psychodynamic therapies such as Emotional Awareness and Expression Therapy (EAET) and Intensive Short Term Psychodynamic Therapy (ISTDP) have recently been evaluated in three systematic reviews and show good results for patients with medically unexplained symptoms. Short-term psychodynamic therapy considers that good treatment outcomes for patients with functional somatic syndromes can be achieved by increasing awareness of emotions and teaching patients to better experience, express and regulate emotions. In several randomized studies, short-term psychodynamic therapy has shown good effects even compared to other treatments, including cognitive behavioral therapy (CBT).

The overall purpose of this research project is to to evaluate psychodynamic emotion-focused interventions (EAET and ISTDP) for patients with medically unexplained symptoms/functional somatic symptoms (MUS/FSD). The project includes several studies that will clarify effects and contribute to information on how care flows in primary care for the patient group can be created.

The research question for this specific study is:

Is internet-based Emotional Awareness and Expression Therapy (I-EAET) with therapist more effective than without therapist support for patients with FSD?

ELIGIBILITY:
Inclusion Criteria:

* The research subject certifies that he/she has undergone medical assessment for his/her physical symptoms.
* The subject rates either moderate distress from bodily symptoms in the PHQ-15 (over 10 points) or severe distress from a single bodily symptom (at least 2 points for this symptom).
* The research participants expresses interest in investigating whether emotional factors such as stress may contribute to symptoms.
* Research subjects either affirm the presence of emotionally difficult life events (affirm at least 1 such event in the Adverse Childhood Experience (ACE-10) or reach the proposed cut-off point of 23p in the PCL-5).
* Drugs used should have been stable for at least 1 month.

Exclusion Criteria:

* Research subjects suffer from ongoing substance abuse (alcohol or drugs) or are deemed to have serious mental illness (psychotic illness, suicidal ideation, antisocial personality disorder etc).
* The research subjects have ongoing medication of a clearly addictive and sedative nature (e.g. benzodiazepines).
* The research subject participates in other psychological treatment focusing on physical symptoms. However, other psychological treatment is allowed where the support therapy does not take place more often than once a month.
* The research subject does not master the Swedish language sufficiently to be able to assimilate written material in Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire -15 (PHQ-15) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings 0-2 on how troublesome somatic symptoms are experienced. Higher scores indicates worse symptom/functioning.
Numeric Rating Scales according to EURONET-SOMA | Change from pre to post treatment (after 10 weeks of treatment)
  Visual analogue scale 0-10 for symptom intensity and symptom interference. Higher scores indicates worse symptom/functioning.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings 0-3 on impact of anxiety symptoms. Higher scores indicates worse symptom/functioning.
Patient Health Questionnaire-9 (PHQ-9) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings 0-3 on impact of depressive symptoms. Higher scores indicates worse symptom/functioning.
Post traumatic stress disorder checklist-5 (PCL-5) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings 0-4 on impact of post traumatic symptoms. Higher scores indicates worse symptom/functioning.
Difficulties in Emotion Regulation Scale-16 (DERS-16) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings on emotional (dys)regulation. Higher scores indicates worse symptom/functioning.
Sheehan Disability Scale (SDS) | Change from pre to post treatment (after 10 weeks of treatment)
  Visual analogue scale 0-10 for symptom interference in daily life. Higher scores indicates worse symptom/functioning.
The revised illness perception questionnaire (IPQ-R) | Change from pre to post treatment (after 10 weeks of treatment)
  Ratings on illness beliefs.

OTHER OUTCOMES:
Mediational measure: DERS-16 | Each week once a week throughout 10 weeks of treatment
  Ratings on emotional (dys)regulation. Higher scores indicates worse symptom/functioning.
Mediational measure: PHQ-15 | Each week once a week throughout 10 weeks of treatment
  Ratings 0-2 on how troublesome somatic symptoms are experienced. Higher scores indicates worse symptom/functioning.
Mediational measure: PHQ-4 | Each week once a week throughout 10 weeks of treatment
  Ratings 0-2 on how troublesome somatic symptoms are experienced. Higher scores indicates worse symptom/functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Original data shared on demand from other researchers and after approval from Swedish Ethical Review Authority.

REFERENCES:
- See also: Information about study project at Stockholm University — https://www.su.se/forskning/forskningsprojekt/k%C3%A4nslofokuserade-digitala-interventioner-f%C3%B6r-patienter-med-medicinskt-of%C3%B6rklarade-symtom